CLINICAL TRIAL: NCT03864120
Title: Understand the Difference Between Clinical Measured Ultrafiltration and Real Ultrafiltration.
Brief Title: Understand the Difference Between Clinical Measured UF and Real UF.
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zanzhe Yu, Principal Investigator, RenJi Hospital
Other Study IDs: 仁济2018（078）
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The importance of ultrafiltration (UF) and fluid status in peritoneal dialysis has been increasingly aware of over the last two decades. There is growing body of observational evidence showing that low UF is related to unfavorable outcome especially in anuric patients. The other side of the problem of UF is excessive fluid removal could volume deplete patients and result in loss of residual renal function and overexposing the membrane to glucose unnecessarily. UF is a double-edged sword. The correct measure of UF is the bottom line of talking about target.

Measuring UF is supposed to be simple and straight forward. The most common way of measuring UF in clinical practice was to weight the effluent bag and minus the manufacture announced fill volume.

Until about 10 years ago, the society first aware that the measurement error in such way is not acceptable. Overfil (the actual volume of dialysate fill in the bag is more than announced) problem was raised from then.

However, there are several other problems around this issue. Firstly, when the product has just been produced overfill is different between manufactory.

Secondly, the overfill volume does change over transportation and storage. But it is not clear how big the change is.

Thirdly, most of the clinics weight the dialysate effluent rather than measure the volume in CAPD, although the specific gravity of dialysate is clearly not going to be 1g/ml.

Taking the fact measuring weight is much easier than measuring volume in CAPD, the question behind is to understand how big the difference is and consequently whether it is acceptable.

All the patients enrolled in the study would be asked to collect all dialysate effluent of the day of their routine peritoneal dialysis adequacy study and bring to the hospital. The exact weight of the bag for PET test (2.5% glucose concentration and dwell time of 4 hour) before and after the dwell and volume measured of the effluent. The dialysate electrolyte, glucose, protein and creatinine level would also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. on PD treatment for at least one month
3. signed the consent

Exclusion Criteria:

1. Peritonitis or recovery from peritonitis for less than one month.
2. On any intra peritoneal treatment apart from peritoneal dialysis.
3. Evidence of decompensated liver cirrhosis or heart failure.
4. Evidence of extra peritoneal leakage, eg. leakage to thoracic cavity, post peritoneal, hernia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18years), both gender, end stage renal disease on PD treatment
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
specific gravity of effluent dialysate is different from water (1g/ml) | For each patient, the outcome would be cross sectional measured at the time the patient does his 6 monthly routine PET test. The data collection time period of the study is 6 month.
  To describe the specific gravity of effluent dialysate, the exact weight and volume of effluent dialysate bags in the standard peritoneal equivalent test (PET, 2.5% glucose concentration, 2L, dwell time 4 hours) dwell would be measured in different patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zanzhe Yu, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Z, Wang Z, Wang Q, Zhang M, Jin H, Ding L, Yan H, Huang J, Jin Y, Davies S, Fang W, Ni Z. Understand the difference between clinical measured ultrafiltrationand real ultrafiltration in peritoneal dialysis. BMC Nephrol. 2021 Nov 15;22(1):382. doi: 10.1186/s12882-021-02589-3. PMID 34781890